CLINICAL TRIAL: NCT05088642
Title: A Phase I Clinical Study Evaluating the Pharmacokinetics and Safety of Hetrombopag Olamine Tablets in Subjects With Mild Hepatic Impairment (Child-Pugh Class A), Moderate Hepatic Impairment (Child-Pugh Class B), and Normal Hepatic Function
Brief Title: A Trial of Hetrombopag in Healthy and Hepatic Impairment Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-109
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Sever Aplastic Anaemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Child-Pugh Class A) (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet
- Moderate hepatic impairment (Child-Pugh Class B) (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet
- Normal hepatic function (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet

INTERVENTIONS:
Drug: Hetrombopag Olamine Tablet — Hetrombopag Olamine Tablet

SUMMARY:
This is a single-dose, open-label, phase I clinical study evaluating the PK of hetrombopag in subjects with mild hepatic impairment (Child-Pugh Class A), subjects with moderate hepatic impairment (Child-Pugh Class B), as well as age-, weight-, and gender-matched subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the study and fully understand the study content, process, and possible adverse reactions; able to complete the study as required by the clinical study protocol;
2. Subjects (and their partners) are willing to adopt effective contraceptive measures from screening to 6 months after the last study administration. See Appendix 1 for specific contraceptive measures;
3. Aged 18-65 years (inclusive), male or female;
4. Body mass index (BMI = weight (kg)/height2 (m2)): 18-30 kg/m2 (inclusive);
5. For subjects with normal hepatic function: normal or abnormal but not clinically significant laboratory findings (hematology, blood biochemistry, urinalysis, and coagulation function);
6. For subjects with normal hepatic function: no history of severe primary disorders involving major organs, including but not limited to the gastrointestinal, respiratory, renal, hepatic, neural, hematological, endocrine, neoplastic, immunological, psychiatric, or cardiovascular and cerebrovascular disorders.

   Subjects with hepatic insufficiency must also meet the following inclusion criteria:
7. Have not received medication within 4 weeks before screening, or have received stable medication for at least 4 weeks for hepatic impairment and/or other concurrent diseases requiring long-term treatment;
8. With Child-Pugh Class A or B hepatic insufficiency caused by prior primary liver disorders (except drug-induced liver diseases).

Exclusion Criteria:

1. Average daily consumption of > 5 cigarettes within 3 months before screening;
2. Allergic constitution, or allergy to any component of hetrombopag olamine tablets;
3. Average daily alcohol consumption of > 15 g for females (e.g., 145 mL of wine, 497 mL of beer, or 43 mL of low-alcohol liquor) and > 25 g for males (e.g., 290 mL of wine, 994 mL of beer, or 86 mL of low-alcohol liquor) within 3 months before screening;
4. History of drug abuse within 3 months before screening;
5. Have donated or lost ≥ 400 mL of blood, or have received blood transfusion within 3 months before screening;
6. Have undergone major surgery within 6 months before screening, or with incomplete healing of surgical incision;
7. History of deep vein thrombosis or other thromboembolic events, or clinical symptoms suggesting thrombophilia;
8. Have received TPO receptor agonists (such as eltrombopag and romiplostim) or TPO within 1 month before screening;
9. Have taken Chinese herbal medicines or any drug that affects the PK of hetrombopag within 14 days before study administration (see Appendix 2 for drug-drug interaction evaluation);
10. Hypertension [systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg, confirmed by a re-measurement];
11. Female subjects who are in lactation or have a positive serum pregnancy test result at screening or during the study;
12. Abnormal and clinically significant 12-lead ECG results (such as tachycardia/bradycardia requiring pharmacological treatment, second- or third-degree atrioventricular block or QTcF interval prolongation (≥ 470 ms for males, ≥ 480 ms for females) (corrected according to Fridericia's formula), or other clinically significant abnormalities assessed by the clinician);
13. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 calculated using the Modification of Diet in Renal Disease (MDRD) equation;
14. Have malignant tumors or history of malignant tumors within 5 years before screening (except treated non-melanoma skin cancer without sign of recurrence and resected cervical intraepithelial neoplasia);
15. For subjects with normal hepatic function: have participated in any drug or medical device clinical trials within 3 months before screening; for subjects with hepatic insufficiency: have participated in any drug or medical device clinical trials within 1 month before screening;
16. For subjects with normal hepatic function: test positive for hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antibody, or syphilis antibody in screening;
17. Probably undergo surgery or be hospitalized during the study;
18. Have consumed alcohol (or positive for breath alcohol test), grapefruit/grapefruit juice, or any food or beverage containing methylxanthine (such as coffee, tea, cola, chocolate, and energy drink), have participated in strenuous physical activities, or have other factors that may affect drug absorption, distribution, metabolism, and excretion within 1 day before study administration;
19. Positive for urine drug screening (morphine or marijuana);
20. Subjects judged by the investigator as unsuitable for participating in this study.

    Additional exclusion criteria for subjects with hepatic insufficiency (those who meet any of the followings are ineligible):
21. History of liver transplant;
22. Liver failure, or liver cirrhosis complicated with hepatic encephalopathy, hepatocellular carcinoma, esophageal and gastric varices hemorrhage, and other complications that, in the opinion of the investigator, make subjects unsuitable for participating in this study;
23. History of any serious diseases, other than primary liver diseases, or history of disorders and/or clinically significant abnormal laboratory findings that, as judged by the investigator, may affect the results of the study, including but not limited to the history of diseases in the circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases.
24. Positive for HIV antibody screening; a rapid plasma reagin (RPR) test is required for a subject who tests positive for syphilis antibodies, and the subject should be excluded if the RPR result is also positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0-120 hours post dose
Area Under the plasma concentration vs time curve (AUC0-120). | 0-120 hours post dose
Area under the blood concentration vs time curve (AUC0-inf). | 0-infinity

SECONDARY OUTCOMES:
Time to Reach Maximum Drug Concentration in Plasma After Single Dose (Tmax) | 0-120 hours post dose
Half-life Associated With the Terminal Slope (t½) | 0-120 hours post dose
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided